CLINICAL TRIAL: NCT05345249
Title: Erector Spinae Plane Block for Reduction of Early Postoperative Pain Scores and Opioid Use in Lumbar Spinal Fusion Surgery, a Prospective Double-blinded Randomized Placebo-controlled Trial
Brief Title: Erector Spinae Plane Block as Pain Management After Lumbar Fusion Surgery
Acronym: RCT-ESPB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ilse van de Wijgert (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Sponsor-Investigator, Ilse van de Wijgert, Principal Investigator, Sint Maartenskliniek
Organization: Sint Maartenskliniek (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0984; 2021-003679-32 (EudraCT Number); NL9640 (Other: Netherlands Trial Register)
Record Dates: First submitted 2022-03-28; First posted 2022-04-25 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Spondylolisthesis; Lumbar Disc Herniation; Lumbar Spinal Stenosis; Lumbar Disc Disease; Lumbar Spondylolisthesis; Lumbar Spondylosis; Lumbar Spine Disease; Lumbar Radiculitis; Spinal Fusion; Fusion of Spine; Spondylosis Lumbosacral Region
Keywords: Erector spinae block; Lumbar interbody fusion; Regional anesthesia; Postoperative pain
MeSH Terms: conditions — Spondylolisthesis; Intervertebral Disc Displacement; Spinal Stenosis; Intervertebral disc disease; Spondylosis; Spinal Diseases; Radiculopathy; Pain, Postoperative | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Patients scheduled for elective lumbar spinal fusion surgery will be studied. Subject of investigation is the locoregional anesthetic technique ESPB. Subjects will be randomized to receive either ESPB with a long-acting local anesthetic or normal saline (placebo). The staff involved (doctors, nurses, OR-personal), as well as the research team and the patient will be blinded for treatment allocation. The study period includes in-hospital time after surgery and follow-up 30 days after surgery. Placement of the ESPB will be performed according to the study protocol, at the end of surgery, after wound closure. The placement of the ESPB is performed according to daily clinical practice as described by Forero et al.
  Postoperative treatment of patients will be according to standard hospital protocol for lumbar spinal fusion surgery.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: After obtaining informed consent, the coordinating researcher creates a study case.
  Patients will be randomly allocated in a 1:1 ratio to either the study group (ESPB) or the control group (placebo) by the hospital's pharmacist on the day of surgery. Permuted block randomization with varying permuted block sizes will be used. This block randomization list will be created by Sealed EnvelopeTM and managed by the hospital's pharmacist. Only the hospital's pharmacist will have access to the randomization list. The staff involved (doctors, nurses, operation room personal), as well as the research team and the patient will be blinded for treatment allocation.
  The hospital's pharmacist prepares the medication on the morning of surgery, delivers it at the operation complex and collects empty syringes after injection in terms of drug accountability.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ESPB with ropivacaine (Experimental): Patients in the experimental group will receive locoregional analgesia via ESPB with injectate consisting of ropivacaine 0.375 mg/mL with no additives, two times 30mL bilaterally at the transverse processs of the T12-vertebra (total dose of 225 mg).
  Interventions: Drug: Ropivacaine Hydrochloride Injection
- ESPB with placebo (Placebo Comparator): Patients in the placebo group will receive an injection performed as the procedure of ESPB with injectate consisting of sodiumchloride 0.9% with no additives, two times 30mL bilaterally at the transverse processs of the T12-vertebra.
  Interventions: Drug: Sodium chloride

INTERVENTIONS:
Drug: Ropivacaine Hydrochloride Injection — Investigating the effectiveness of erector spinae plane block with ropivacaine for lumbar spinal fusion surgery versus placebo.
  Other Names: SMPC h104944; Ropivacaine HCl
  Arms: ESPB with ropivacaine
Drug: Sodium chloride — Placebo comparator
  Other Names: SMPC h55227; NaCl 0.9%
  Arms: ESPB with placebo

SUMMARY:
Rationale: Lumbar spine surgery is associated with high postoperative pain scores and analgesic use, despite use of multimodal analgesia. The erector spinae plane block (ESPB) is a promising locoregional anesthetic technique for this type of surgery. The literature is not yet conclusive about the effectiveness of this technique on reducing postoperative pain intensity.

Objective: The objective of this study is to evaluate the analgesic effect of ESPB as add-on therapy to multimodal analgesia on early postoperative pain intensity after lumbar spinal fusion surgery compared to placebo.

Study design: The study is designed as a prospective mono-centre, randomized, double-blinded, placebo-controlled trial.

Study population: 76 patients ≥ 18 years of age requiring elective lumbar spinal fusion surgery involving one to four fusion levels.

Intervention: Patients will receive ultrasound-guided ESPB with either ropivacaine or placebo at the end of surgery.

Main study parameters/endpoints: Main study parameter is pain intensity upon emergence from anesthesia measured with the Numeric Rating Scale. A minimal clinically important difference is considered to be a decrease of 1.5 points. Secondary endpoints are pain intensity during hospital stay and after 30 days, opioid use during hospital stay and after 30 days, opioid side effects, use of anti-emetics, time to first opioid use/request, length of hospital stay, quality of recovery at discharge.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The Sint Maartenskliniek is experienced in applying locoregional analgesia, the use of ropivacaine and using sonography. The procedure of administering ESPB has a very low risk of complications. Receiving placebo is justifiable because this group will not be withhold standard treatment. The risks of receiving placebo are negligible. The patients will visit the clinic at regular follow-up moments.

DETAILED DESCRIPTION:
Rationale: Lumbar spine surgery is associated with high postoperative pain scores and analgesic use. Despite multimodal pain treatment, time to first rescue treatment with opioids is often short and necessary on the Post Anesthesia Care Unit (PACU). Latest scientific insights show most pain interventions produce mild analgesic effects, and advise a multimodal regimen based upon systemic analgesics consisting of at least gabapentoids, ketamine and opioids. Therefore, in our clinic (Sint Maartenskliniek, Nijmegen, the Netherlands), multimodal analgesia in spine surgery is now gold standard, with opioids as first choice postoperative rescue treatment. However, despite multimodal treatment, patients who underwent lumbar spine surgery still develop severe postoperative pain.

A different possible measure to lower the risk of postoperative pain is locoregional anesthesia. The Sint Maartenskliniek has a long history of applying locoregional anesthesia in orthopedic surgery. Locoregional anesthesia provides effective analgesia without systemic side-effects like drowsiness or nausea, thereby reducing perioperative systemic drug use and possibly reducing the risk of persistent postsurgical pain. A novel locoregional anesthetic technique is the erector spinae plane block (ESPB). Good quality evidence exists for the effectiveness of this technique in breast cancer surgery and video assisted thoracoscopy (VATS). Although ESPB seems a promising analgesic technique for lumbar spine surgery patients not responding to the multimodal pain treatment regimen, sufficient high quality evidence is lacking. A recent systematic review summarized the evidence of ESPB for lumbar spine surgery, including two randomized clinical trials (RCT), showing beginning evidence of reduced postoperative opioid consumption and decreased pain scores. However, these trials contained a small sample size, were not blinded or lacked a comparator. Furthermore, little information on postoperative hospital stay is provided. This results in ESPB not being widely accepted in lumbar spine surgery. The larger, double-blinded, placebo-controlled methodology in this proposed trial aims to contribute to the scientific evidence for the effectiveness of EPSB in a multimodal analgesia management setting.

Objective: The primary objective of the study is to evaluate the analgesic effect of ESPB on early postoperative pain after lumbar spinal fusion surgery. Therefore the pain intensity in the postoperative care unit upon emergence, using the Numeric Rating Scale (NRS) for pain, will be the primary outcome parameter of this study. The null hypothesis states there is no difference in effectiveness of the ESPB compared to placebo on early postoperative pain intensity measured with NRS in patients that underwent lumbar spinal fusion surgery. This hypothesis will be tested two-sided, with α = 0.05.

Study design: This study is designed as a prospective, mono-center, double-blinded, randomized, placebo controlled trial. The study will be performed at the Sint Maartenskliniek, Nijmegen, the Netherlands. The study will be performed in accordance with the ICH E6(R1) Good Clinical Practice (GCP) guidelines. The duration of the study will be determined according to the progress of inclusion. Patients scheduled for elective lumbar spinal fusion surgery will be studied. Subject of investigation is the locoregional anesthetic technique ESPB. Subjects will be randomized to receive either ESPB with a long-acting local anesthetic or normal saline (placebo).

The staff involved (doctors, nurses, OR-personal), as well as the research team and the patient will be blinded for treatment allocation. The study period includes in-hospital time after surgery and follow-up 30 days after surgery. Placement of the ESPB will be performed according to the study protocol, at the end of surgery, after wound closure. The placement of the ESPB is performed according to daily clinical practice as described by Forero et al. Postoperative treatment of patients will be according to standard hospital protocol for lumbar spinal fusion surgery.

Study population: 76 patients undergoing elective lumbar spinal fusion surgery involving one to four fusion levels will be recruited.

Main study parameters/endpoints: Main study parameter is pain intensity upon emergence from anesthesia measured with the Numeric Rating Scale. A minimal clinically important difference is considered to be a decrease of 1.5 points. Secondary endpoints are pain intensity during hospital stay and after 30 days, opioid use during hospital stay and after 30 days, opioid side effects, use of anti-emetics, time to first opioid use/request, length of hospital stay, quality of recovery at discharge.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The Sint Maartenskliniek is experienced in applying locoregional analgesia, the use of ropivacaine and using sonography. The procedure of administering ESPB has a very low risk of complications. Receiving placebo is justifiable because this group will not be withhold standard treatment. The risks of receiving placebo are negligible. The patients will visit the clinic at regular follow-up moments.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Patients planned for elective lumbar spinal fusion surgery with a dorsal surgical approach;
* 1-4 fusion level spine surgery;
* Written informed consent.

Exclusion Criteria:

* A Body Mass Index (BMI) > 40 kg/m²;
* ASA physical health classification > 3;
* Patients who will undergo spine surgery involving less than 2 or more than 4 levels of fusion, scoliosis surgery*;
* Patients who will undergo circumferent spine surgery;
* Patients with an active, local infection or systemic infection;
* Patients with an allergy to one or more medications used in the study;
* Patients with any contraindication to a regional anesthetic technique;
* Kidney- or liver failure inhibiting the systemic use of paracetamol and/or NSAIDs;
* Acute surgeries;
* Patients with a history of drugs or alcohol abuse;
* Pregnancy;
* Cognitive impairment;
* Inability to speak or understand the Dutch language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
Pain intensity one hour after arrival at post-anesthesia care unit | 1 hour after arrival at PACU
  Numeric Rating Scale (NRS) for pain 0-10 (0 = no pain, 10 = maximum pain) as asked by PACU-nurse

SECONDARY OUTCOMES:
Acceptability of pain | 1 hour after arrival at PACU
  Yes/no
Opioid use | 0-12 hours, 12-24 hours after surgery
  total morphine equivalent dose as extracted from the electronic medical file and PCIA pump
Presence of opioid side effects | 12 hours, 24 hours after surgery
  Nausea, vomiting and use of anti-emetics as documented in electronic medical file
Time to first opioid use/request | 12 hours after surgery
  defined as minutes
Time to first mobilization | 72 hours after surgery
  defined as hours
Length of hospital stay | up to 30 days after surgery
  defined as days
Pain intensity | on postoperative admission days, 30 days
  Numeric Rating Scale (NRS) for pain 0-10 (0 = no pain, 10 = maximum pain)
Opioid use | 30 days after surgery
  Do you use opioids yes/no
Quality of recovery | Postoperative day 1 and 3
  Quality of Recovery-15 questionnaire (Dutch version). Score 0-150 (0 = worst recovery, 150 = perfect recovery)
Adverse events | 0-30 days after surgery
  (Serious) adverse events during study period

OTHER OUTCOMES:
Drain wound leakage | Postoperative day 1, 2 and 3
  mLs of drain wound leakage, if drain is present

CONTACTS AND LOCATIONS:
Overall Officials: M.G.E. Fenten, MSc, PhD, MD, Principal Investigator — Sint Maartenskliniek
Locations (1):
- Sint Maartenskliniek, Ubbergen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
DANS EASY will be data repository for open access.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After end of inclusion period for at least 5 years.
Access Criteria: DANS EASY will be data repository for open access. FAIR Guiding Principles are followed to make data Findable, Accessible, Interoperable and Reusable. An Open Access-licence is required to consult the data.
URL: https://dans.knaw.nl/en/data-services/easy/

REFERENCES:
- [Background] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233
- [Background] Alboog A, Bae S, Chui J. Anesthetic management of complex spine surgery in adult patients: a review based on outcome evidence. Curr Opin Anaesthesiol. 2019 Oct;32(5):600-608. doi: 10.1097/ACO.0000000000000765. PMID 31461735
- [Background] Huang W, Wang W, Xie W, Chen Z, Liu Y. Erector spinae plane block for postoperative analgesia in breast and thoracic surgery: A systematic review and meta-analysis. J Clin Anesth. 2020 Nov;66:109900. doi: 10.1016/j.jclinane.2020.109900. Epub 2020 Jun 2. PMID 32502778
- [Background] Qiu Y, Zhang TJ, Hua Z. Erector Spinae Plane Block for Lumbar Spinal Surgery: A Systematic Review. J Pain Res. 2020 Jul 1;13:1611-1619. doi: 10.2147/JPR.S256205. eCollection 2020. PMID 32669870
- [Background] Yayik AM, Cesur S, Ozturk F, Ahiskalioglu A, Ay AN, Celik EC, Karaavci NC. Postoperative Analgesic Efficacy of the Ultrasound-Guided Erector Spinae Plane Block in Patients Undergoing Lumbar Spinal Decompression Surgery: A Randomized Controlled Study. World Neurosurg. 2019 Jun;126:e779-e785. doi: 10.1016/j.wneu.2019.02.149. Epub 2019 Mar 8. PMID 30853517
- [Background] Singh S, Choudhary NK, Lalin D, Verma VK. Bilateral Ultrasound-guided Erector Spinae Plane Block for Postoperative Analgesia in Lumbar Spine Surgery: A Randomized Control Trial. J Neurosurg Anesthesiol. 2020 Oct;32(4):330-334. doi: 10.1097/ANA.0000000000000603. PMID 31033625
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/49/NCT05345249/Prot_SAP_000.pdf